CLINICAL TRIAL: NCT03089125
Title: Brief Behavioral Intervention for Dyspnea in Patients With Advanced Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Joseph A. Greer, Ph.D., Associate Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-476
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Nurse administered dyspnea intervention
Who Masked: Outcomes Assessor
Masking Description: Research staff collecting patient-reported measures will be blind to study assignment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patients will receive any usual care for their dyspnea as deemed appropriate by their clinicians.
  Interventions: Other: Usual Care
- Dyspnea Intervention (Experimental): Dyspnea intervention will be administered over two sessions
  Patients will receive:
  * Psychoeducation
  * Relaxation training for reducing physiological stress
  * Behavioral techniques for managing acute breathlessness
  Interventions: Behavioral: Dyspnea Intervention; Other: Usual Care

INTERVENTIONS:
Behavioral: Dyspnea Intervention — Dyspnea intervention will be administered over two sessions
  Patients will receive:
  * Psychoeducation
  * Relaxation training for reducing physiological stress
  * Behavioral techniques for managing acute breathlessness
  Arms: Dyspnea Intervention
Other: Usual Care — Patients will receive any usual care for their dyspnea as deemed appropriate by their clinicians

SUMMARY:
This research study is evaluating a behavioral intervention designed to help people with advanced lung cancer manage dyspnea (i.e., breathlessness or shortness-of-breath).

DETAILED DESCRIPTION:
Many individuals with advanced lung cancer experience debilitating breathlessness at some point during the course of their illness. Unfortunately, few interventions exist to treat this distressing symptom of cancer.

The purpose of this study is to test the efficacy of a brief behavioral intervention may help relieve breathlessness in individuals with advanced lung cancer. Participants will have a 50/50 chance of receiving the behavioral intervention or standard care. The principal investigator of the study, Dr. Joseph Greer, is a licensed clinical psychologist who has trained oncology nurses in how to deliver the behavioral intervention. The oncology nurses will meet with participants during their outpatient oncology appointments, such as chemotherapy infusions, to review the behavioral skills that may help with breathlessness. This intervention involves no medications but rather teaches patients skills for breathing control and relaxation of the body.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of either NSCLC, SCLC, or mesothelioma, not being treated with curative intent
* Self-reported shortness of breath (a score of 2 or greater on the Modified Medical Research Council Dyspnea Scale)
* Eastern Cooperative Oncology Group (ECOG) Performance Status from 0 (asymptomatic) to 2 (symptomatic and in bed <50% of day)
* The ability to read and respond to questions English
* Primary cancer care at the Massachusetts General Hospital (MGH) Cancer Center or Dana-Farber Cancer Institute (DFCI)
* Age >18 years

Exclusion Criteria:

* Cognitive or psychiatric conditions prohibiting study consent or participation.
* A treating clinician who reports that the patient is inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Greer, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greer JA, Post KE, Chabria R, Aribindi S, Brennan N, Eche-Ugwu IJ, Halpenny B, Fox E, Lo S, Waldman LP, Pintro K, Rabideau DJ, Pirl WF, Cooley ME, Temel JS. Randomized Controlled Trial of a Nurse-Led Brief Behavioral Intervention for Dyspnea in Patients With Advanced Lung Cancer. J Clin Oncol. 2024 Oct 20;42(30):3570-3580. doi: 10.1200/JCO.24.00048. Epub 2024 Aug 1. PMID 39088766

RESULTS

PARTICIPANT FLOW:
Groups:
- Dyspnea Intervention: Dyspnea intervention will be administered over two sessions
  Patients will receive:
  * Psychoeducation
  * Relaxation training for reducing physiological stress
  * Behavioral techniques for managing acute breathlessness
  Dyspnea Intervention: Dyspnea intervention will be administered over two sessions
  Patients will receive:
  * Psychoeducation
  * Relaxation training for reducing physiological stress
  * Behavioral techniques for managing acute breathlessness
  Usual Care: Patients will receive any usual care for their dyspnea as deemed appropriate by their clinicians
Period: Overall Study
Arm/Group | Usual Care | Dyspnea Intervention
Started | 121 | 126
Completed | 99 | 94
Not Completed | 22 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Dyspnea Intervention | Total
Number analyzed (Participants) | 121 | 126 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.44 (10.08) | 66.83 (11.47) | 66.15 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 68 | 138
  Male | 51 | 58 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 118 | 117 | 235
  Unknown or Not Reported | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 113 | 110 | 223
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 121 | 126 | 247
Modified Medical Research Council Dyspnea Scale (mMRCDS) [Mean (Standard Deviation); unit: units on a scale] — The Modified Medical Research Council Dyspnea Scale evaluates dyspnea-related functional impairment. Total scale score range: 0 (minimum) to 4 (maximum), with higher scores indicating worse dyspnea.
  units on a scale | 2.60 (0.75) | 2.59 (0.72) | 2.60 (0.73)
Cancer Dyspnoea Scale (CDS) [Mean (Standard Deviation); unit: units on a scale] — The Cancer Dyspnoea Scale assesses dyspnea-related effort, anxiety, and physical discomfort. Total scale score range: 0 (minimum) to 48 (maximum), with higher scores indicating worse dyspnea.
  units on a scale | 12.61 (7.51) | 11.13 (6.51) | 11.85 (7.05)
Functional Assessment of Cancer Therapy - Lung (FACT-L) [Mean (Standard Deviation); unit: units on a scale] — The Functional Assessment of Cancer Therapy - Lung Scale measures overall quality of life, including physical, social, emotional, and functional wellbeing as well as lung cancer-specific symptoms. Total scale score range: 0 (minimum) to 136 (maximum), with higher scores indicating better quality of life.
  units on a scale | 87.23 (16.36) | 90.19 (18.59) | 88.74 (17.56)
Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale - Anxiety Subscale assesses anxiety symptoms in the past week. Total subscale score range: 0 (minimum) to 21 (maximum), with higher scores indicating worse anxiety symptoms.
  units on a scale | 6.68 (3.76) | 5.37 (3.80) | 6.01 (3.83)
Hospital Anxiety and Depression Scale (HADS) - Depression Subscale [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale - Depression Subscale assesses depression symptoms in the past week. Total subscale score range: 0 (minimum) to 21 (maximum), with higher scores indicating worse depression symptoms.
  units on a scale | 6.40 (3.16) | 5.73 (3.72) | 6.06 (3.47)
Godin-Shephard Leisure Time Physical Activity Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Godin-Shephard Leisure Time Physical Activity Questionnaire assesses the frequency and extent of physical activity over the course of one week. Total scale score range: 0 (minimum; insufficiently active) to 24 or greater (maximum; active), with higher scores indicating greater physical activity. Population: 6 participants in the Usual Care Group and 9 participants in the Dyspnea Intervention Group did not complete the baseline Godin-Shephard Leisure Time Physical Activity Questionnaire.
  units on a scale
    number analyzed (Participants) | 115 | 117 | 232
    (all) | 11.19 (18.20) | 12.29 (16.91) | 11.75 (17.53)
Actigraphy [Mean (Standard Deviation); unit: Percent time spent immobile while awake] — Participants were asked to wear a wrist actigraph device during a consecutive 3-day period at baseline and again at week 8 (primary outcome time point). Percentages (0-100%) represent proportion of time spent immobile while awake. Population: 37 participants in the Usual Care Group and 37 participants in the Dyspnea Intervention Group did not have three consecutive days of actigraphy data at baseline.
  Percent time spent immobile while awake
    number analyzed (Participants) | 84 | 89 | 173
    (all) | 50.48 (13.62) | 47.61 (11.19) | 49.00 (12.48)

OUTCOME MEASURES:

1. Primary Outcome: Modified Medical Research Council Dyspnea Scale (mMRCDS)
Description: Compare the difference between study groups in the Modified Medical Research Council Dyspnea Scale severity score at 8 weeks. The Modified Medical Research Council Dyspnea Scale scores range from 0 (minimum) to 4 (maximum), with higher scores indicating more severe dyspnea.
Time Frame: 8 weeks
Population: Reasons for missing data include participants being unable to complete study measures due to worsening illness or death, withdrawing from the study, declining to complete the measures, or being lost to follow-up or transferring care.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 98 | 92
units on a scale | 1.88 [1.69 to 2.07] | 1.55 [1.35 to 1.75]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.038, ANCOVA — Bonferroni-adjusted P-value; ANCOVA models control for cancer type, study site, and baseline scores of outcome variable; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.61 to -0.05]

2. Primary Outcome: Cancer Dyspnoea Scale (CDS)
Description: Compare the difference between study groups in the Cancer Dyspnoea Scale scores at 8 weeks. The Cancer Dyspnoea Scale scores range from 0 (minimum) to 48 (maximum), with higher scores indicating worse dyspnea.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 99 | 92
units on a scale | 10.01 [8.87 to 11.15] | 9.47 [8.28 to 10.65]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p > 0.99, ANCOVA — Bonferroni-adjusted P-value; ANCOVA models control for cancer type, study site, and baseline scores of outcome variable; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-2.20 to 1.10]

3. Secondary Outcome: Functional Assessment of Cancer Therapy - Lung (FACT-L)
Description: Compare the difference between study groups in the Functional Assessment of Cancer Therapy - Lung Scale scores at 8 weeks. The Functional Assessment of Cancer Therapy - Lung Scale scores range from 0 (minimum) to 136 (maximum), with higher scores indicating better quality of life.
Time Frame: 8 weeks
Population: Reasons for missing data include participants being unable to complete study measures due to worsening illness or death, withdrawing from the study, declining to complete the measures, or being lost to follow-up or transferring their care to another institution.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 97 | 91
units on a scale | 91.40 [88.91 to 93.89] | 93.00 [90.43 to 95.57]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.380, ANCOVA; ANCOVA models control for cancer type, study site, and baseline scores of outcome variable; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [-1.98 to 5.18]

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale
Description: Compare the difference between study groups in the Hospital Anxiety and Depression Scale - Anxiety Subscale scores at 8 weeks. The Hospital Anxiety and Depression Scale - Anxiety Subscale scores range from 0 (minimum) to 21 (maximum), with higher scores indicating worse anxiety symptoms.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 99 | 92
units on a scale | 5.85 [5.27 to 6.42] | 5.84 [5.25 to 6.43]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.990, ANCOVA; ANCOVA models control for cancer type, study site, and baseline scores of outcome variable; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.83 to 0.82]

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Depression Subscale
Description: Compare the difference between study groups in the Hospital Anxiety and Depression Scale - Depression Subscale scores at 8 weeks. The Hospital Anxiety and Depression Scale - Depression Subscale scores range from 0 (minimum) to 21 (maximum), with higher scores indicating worse depression symptoms.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 99 | 92
units on a scale | 6.09 [5.50 to 6.67] | 5.59 [4.99 to 6.20]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.251, ANCOVA; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.34 to 0.35]

6. Secondary Outcome: Activity Level (Self-report: Godin-Shephard Leisure Time Physical Activity Questionnaire)
Description: Compare the difference between study groups in the Godin-Shephard Leisure Time Physical Activity Questionnaire scores at 8 weeks. The Godin-Shephard Leisure Time Physical Activity Questionnaire is a 4-item measure that assesses the frequency and extent of physical activity during free time over the course of one week, with scores ranging from 0 (minimum; insufficiently active) to 24 or greater (maximum; active), with higher scores indicating greater physical activity.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 90 | 74
units on a scale | 12.73 [8.43 to 17.03] | 11.24 [6.50 to 15.98]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.647, ANCOVA; ANCOVA models control for cancer type, study site, and baseline scores of outcome variable; Mean Difference (Final Values) = -1.49, 95% CI 2-sided [-7.90 to 4.92]

7. Secondary Outcome: Activity Level (Objective Measure: Actigraphy)
Description: Compare the difference between study groups in the percentage of time spent immobile but awake over a consecutive three day period per actigraphy at 8 weeks. Scores range from 0% to 100%, with higher scores indicating a greater percentage of time spent immobile while awake over a consecutive three day period.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percent time spent immobile while awake
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 55 | 47
percent time spent immobile while awake | 45.80 [43.06 to 48.53] | 47.42 [44.46 to 50.38]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.431, ANCOVA — ANCOVA models control for cancer type, study site, and baseline scores of outcome variable; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [-2.45 to 5.71]

8. Other Pre Specified Outcome: Modified Medical Research Council Dyspnea Scale (mMRCDS)
Description: Compare the difference between study groups in the estimated slopes of the scores on the Modified Medical Research Council Dyspnea Scale over all four assessment timepoints of 8-week intervals (i.e., baseline, 8 weeks, 16 weeks, and 24 weeks) using linear mixed effects models. The Modified Medical Research Council Dyspnea Scale scores range from 0 (minimum) to 4 (maximum), with higher scores indicating more severe dyspnea.
Time Frame: 24 weeks
Population: The analysis sample includes the total number of participants by group who completed at least one Modified Medical Research Council Dyspnea Scale outcome measure from baseline to 24 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: mean change in scores on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 121 | 126
mean change in scores on a scale | -0.89 [-1.16 to -0.61] | -0.95 [-1.24 to -0.66]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.710, Mixed Models Analysis; Estimated between-group difference in change in scores per every 8 weeks from baseline through week 24, controlling for cancer type and study site; Between-group diff in change per 8 weeks = -0.06, 95% CI 2-sided [-0.38 to 0.26]

9. Other Pre Specified Outcome: Cancer Dyspnoea Scale (CDS)
Description: Compare the difference between study groups in the estimated slopes of the scores on the Cancer Dyspnoea Scale over all four assessment timepoints of 8-week intervals (i.e., baseline, 8 weeks, 16 weeks, and 24 weeks) using linear mixed effects models. The Cancer Dyspnoea Scale scores range from 0 (minimum) to 48 (maximum), with higher scores indicating worse dyspnea.
Time Frame: 24 weeks
Population: The analysis sample includes the total number of participants by group who completed at least one Cancer Dyspnoea Scale outcome measure from baseline to 24 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: mean change in scores on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 121 | 126
mean change in scores on a scale | -2.63 [-4.13 to -1.13] | -2.26 [-3.84 to -0.67]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.677, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Between-group diff in change per 8 weeks = 0.38, 95% CI 2-sided [-1.40 to 2.16]

10. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy - Lung (FACT-L)
Description: Compare the difference between study groups in the estimated slopes of the scores on the Functional Assessment of Cancer Therapy - Lung Scale over all four assessment timepoints of 8-week intervals (i.e., baseline, 8 weeks, 16 weeks, and 24 weeks) using linear mixed effects models. The Functional Assessment of Cancer Therapy - Lung Scale scores range from 0 (minimum) to 136 (maximum), with higher scores indicating better quality of life.
Time Frame: 24 weeks
Population: The analysis sample includes the total number of participants by group who completed at least one Functional Assessment of Cancer Therapy - Lung Scale outcome measure from baseline to 24 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: mean change in scores on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 121 | 126
mean change in scores on a scale | 4.86 [1.57 to 8.14] | 2.91 [-0.60 to 6.41]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.330, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Between-group diff in change per 8 weeks = -1.95, 95% CI 2-sided [-5.87 to 1.97]

11. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale
Description: Compare the difference between study groups in the estimated slopes of the scores on the Hospital Anxiety and Depression Scale - Anxiety Subscale over all four assessment timepoints of 8-week intervals (i.e., baseline, 8 weeks, 16 weeks, and 24 weeks) using linear mixed effects models. The Hospital Anxiety and Depression Scale - Anxiety Subscale scores range from 0 (minimum) to 21 (maximum), with higher scores indicating worse anxiety symptoms.
Time Frame: 24 weeks
Population: The analysis sample includes the total number of participants by group who completed at least one Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale outcome measure from baseline to 24 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: mean change in scores on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 121 | 126
mean change in scores on a scale | -1.00 [-1.73 to -0.28] | -0.28 [-1.04 to 0.49]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.098, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Between-group diff in change per 8 weeks = 0.73, 95% CI 2-sided [-0.13 to 1.59]

12. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale (HADS) - Depression Subscale
Description: Compare the difference between study groups in the estimated slopes of the scores on the Hospital Anxiety and Depression Scale - Depression Subscale over all four assessment timepoints of 8-week intervals (i.e., baseline, 8 weeks, 16 weeks, and 24 weeks) using linear mixed effects models. The Hospital Anxiety and Depression Scale - Depression Subscale scores range from 0 (minimum) to 21 (maximum), with higher scores indicating worse depression symptoms.
Time Frame: 24 weeks
Population: The analysis sample includes the total number of participants by group who completed at least one Hospital Anxiety and Depression Scale - Depression Subscale outcome measure from baseline to 24 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: mean change in scores on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 121 | 126
mean change in scores on a scale | -0.18 [-0.89 to 0.53] | -0.10 [-0.85 to 0.66]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.845, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Between-group diff in change per 8 weeks = 0.08, 95% CI 2-sided [-0.76 to 0.93]

13. Other Pre Specified Outcome: Activity Level (Self-report: Godin-Shephard Leisure Time Physical Activity Questionnaire)
Description: Compare the difference between study groups in the estimated slopes of the scores on the Godin-Shephard Leisure Time Physical Activity Questionnaire over all four assessment timepoints of 8-week intervals (i.e., baseline, 8 weeks, 16 weeks, and 24 weeks) using linear mixed effects models. The Godin-Shephard Leisure Time Physical Activity Questionnaire is a 4-item measure that assesses the frequency and extent of physical activity during free time over the course of one week, with scores ranging from 0 (minimum; insufficiently active) to 24 or greater (maximum; active), with higher scores indicating greater physical activity.
Time Frame: 24 weeks
Population: The analysis sample includes the total number of participants by group who completed at least one Godin-Shephard Leisure Time Physical Activity Questionnaire outcome measure from baseline to 24 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: mean change in scores on a scale
Arm/Group | Usual Care | Dyspnea Intervention
Number analyzed (Participants) | 119 | 121
mean change in scores on a scale | 0.54 [-5.30 to 6.38] | 1.28 [-5.09 to 7.65]
Statistical Analysis 1: Comparison: Usual Care vs Dyspnea Intervention; Test type: Superiority; p = 0.837, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Between-group diff in change per 8 weeks = 0.74, 95% CI 2-sided [-6.33 to 7.77]

14. Other Pre Specified Outcome: Examine Potential Mediators of Intervention Effects on Patient-reported Outcomes
Description: Examine the degree to which intervention effects on patient reported outcomes are mediated by improved mastery in managing breathlessness (as measured by the Chronic Respiratory Disease Questionnaire)
Time Frame: 24 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Examine Potential Moderators of Intervention Effects on Dyspnea
Description: Examine whether differences in reported dyspnea are moderated by patient demographic and clinical factors
Time Frame: 24 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Health Service Utilization
Description: Examine differences between study groups in rates of emergency department and hospitalizations
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment (baseline) through 24 weeks.
Arm/Group | Usual Care | Dyspnea Intervention
All-Cause Mortality (participants affected / at risk) | 23/121 | 17/126
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/126
Other Adverse Events (participants affected / at risk) | 0/121 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT03089125/Prot_SAP_000.pdf